CLINICAL TRIAL: NCT04056208
Title: The Effect of Pistachios on Risk Factors for Cardiometabolic Disease in Individuals With Pre-diabetes: a Randomized, Cross-over Study
Brief Title: Pistachios Blood Sugar Control, Heart and Gut Health
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PKE Pistachio
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Crossover assignment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evening Pistachio Consumption (Active Comparator): Participants will consume two ounces per day (57 g) of pistachios as an evening snack (i.e., after dinner and before sleep).
  Interventions: Drug: Pistachio
- Usual care (Active Comparator): Advice to consume a snack that contains 1-2 exchanges (15-30 g of carbohydrate) as an evening snack - this is consistent with the current standard of care for people with impaired fasting glucose.
  Interventions: Other: Usual care

INTERVENTIONS:
Drug: Pistachio — Unsalted pistachios
  Arms: Evening Pistachio Consumption
Other: Usual care — Advice and resources will be provided
  Arms: Usual care

SUMMARY:
A two-period randomized crossover study will be conducted to evaluate the effect of nighttime pistachio consumption (i.e., after dinner and before sleep) on fasting blood sugar levels, longer-term blood sugar control, and risk factors for heart disease. This study will also investigate how pistachios affects gut health.

DETAILED DESCRIPTION:
A two-period randomized crossover trial will be conducted. Participants will be randomized to receive each treatment for 12 weeks followed by a minimum 4-week wash-out period. During the pistachio treatment, participants will consume two ounces per day (57 g) of pistachios as an evening snack. During the control phase subjects will be given advice to consume 1-2 exchanges of carbohydrate as an evening snack, which is consistent with usual care. Markers of glycemic control, cardiovascular risk factors and gut health will be assessed at the beginning and the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥25 and ≤45 kg/m2
* Fasting plasma glucose 100 - 125 mg/dL
* non-Smoking

Exclusion Criteria:

* Diagnosed diabetes or fasting glucose >126 mg/dl
* Systolic blood pressure >160mmHg or diastolic blood pressure >100mmHg)
* Prescribed anti-hypertensive, lipid lowering or glucose lowering drugs
* Established cardiovascular disease, stroke, diabetes, liver, kidney or autoimmune disease or inflammatory conditions
* Use of supplements (psyllium, fish oil, soy lecithin, phytoestrogens) and botanicals and not willing to cease for the duration of the study
* Women who are pregnant, lactating, planning to become pregnant or have given birth in the past year
* Weight loss of >=10% of body weight within the 6 months prior to enrolling in the study
* Smoking or use of any tobacco products
* Allergy/intolerance/sensitive to pistachios
* Consumption of >14 alcoholic drinks/week
* Shift-workers and those who cannot consume a snack in the evening

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Fasting plasma glucose concentration | 12 weeks
  Fasting blood glucose (mg/dL)

SECONDARY OUTCOMES:
HbA1c | 12 weeks
  HbA1c (%) will be assessed at the beginning and end of each treatment period
Serum insulin concentration (mIU/L) | 12 weeks
  fasting serum insulin levels assessed by blood draw
Peripheral systolic and diastolic blood pressure (mm Hg) | 12 weeks
  Blood pressure measured assessed using a SphymoCor Xcel (Atcor Medical).
Central systolic and diastolic blood pressure (mm Hg) | 12 weeks
  Blood pressure measured assessed using a SphymoCor Xcel (Atcor Medical).
Carotid-femoral pulse wave velocity (m/s) | 12 weeks
  A measure of arterial stiffness assessed using a SphymoCor Xcel (Atcor Medical). A higher percentage value is indicative of greater arterial stiffness.
Augmentation Index (%) | 12 weeks
  A measure of arterial stiffness assessed using a SphymoCor Xcel (Atcor Medical). A higher percentage value is indicative of greater arterial stiffness.
LDL cholesterol concentration (mg/dL) | 12 weeks
  Assessed using fasting blood draw
HDL cholesterol concentration | 12 weeks
  Assessed using fasting blood draw
Total cholesterol concentration | 12 weeks
  Assessed using fasting blood draw
Triglyceride concentration | 12 weeks
  Assessed using fasting blood draw
HOMA-IR | 12 weeks
  Assessed using fasting blood draw and standardized HOMA-IR calculation. Fasting plasma glucose multiplied by fasting plasma insulin divided by 405.
waist circumference (cm) | 12 weeks
  Measured 10 cm above the navel
body weight (lbs) | 12 weeks
  Assessed using calibrated scale in Clinical Research Center
Diet quality: Healthy Eating Index 2015 | 12 weeks
  Assessed using the Healthy Eating Index 2015
Change in the composition of the gut microbiome | 12 weeks
  microbiome composition assessed using fecal collection kit

CONTACTS AND LOCATIONS:
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riley TM, Wright J, Lamendella R, Bisanz JE, Chen See J, Kanani K, Kris-Etherton PM, Petersen KS. Nighttime Pistachio Consumption Alters Stool Microbiota Diversity and Taxa Abundance Compared with Education to Consume 1-2 Carbohydrate Exchanges (15-30 grams) over 12 Weeks in Adults with Prediabetes: A Secondary Analysis from a Randomized Crossover Trial. Curr Dev Nutr. 2025 May 27;9(7):107481. doi: 10.1016/j.cdnut.2025.107481. eCollection 2025 Jul. PMID 40612050
- [Derived] Riley TM, Kris-Etherton PM, Hart TL, Petersen KS. Intake of Pistachios as a Nighttime Snack Has Similar Effects on Short- and Longer-Term Glycemic Control Compared with Education to Consume 1-2 Carbohydrate Exchanges in Adults with Prediabetes: A 12-Wk Randomized Crossover Trial. J Nutr. 2024 Apr;154(4):1219-1231. doi: 10.1016/j.tjnut.2024.01.021. Epub 2024 Jan 24. PMID 38278217